CLINICAL TRIAL: NCT05907512
Title: The Safety and Efficacy of Endostar Combined With Toripalimab as Postoperative Adjuvant Therapy for Resectable Stage III-Oligometastatic Stage IV Cutaneous Melanoma: A Prospective, Single-arm, Open-label, Phase II Clinical Study
Brief Title: Endostar Plus Toripalimab as Adjuvant Therapy for Resectable Stage III-Oligometastatic Stage IV Cutaneous Melanoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Chunmeng Wang, Dr. & Prof., Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20009224-4-2304B
Record Dates: First submitted 2023-06-08; First posted 2023-06-18 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Clinical Stage III Cutaneous Melanoma AJCC v8; Clinical Stage IV Cutaneous Melanoma AJCC v8
Keywords: Melanoma; Stage III-oligometastatic IV; Endostar; Toripalimab; Combination therapy
MeSH Terms: conditions — Melanoma | interventions — endostar protein; toripalimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Drug group (Experimental)
  Interventions: Drug: Endostar; Drug: Toripalimab

INTERVENTIONS:
Drug: Endostar — The dose of 210 mg (14 vials) is administered by intravenous pump from Day 1 to Day 3 of each course, every 4 weeks as a cycle, until disease recurrence, metastasis or intolerable toxicity, and up to 6 courses of administration.
Drug: Toripalimab — 3 mg/kg by intravenous drip every 2 weeks (Day 1 and Day 15 of each cycle) in a 4-week cycle until disease recurrence, metastasis, or intolerable toxicity for up to 1 year (about 13 cycles).

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of Endostar combined with Toripalimab in the adjuvant treatment of resectable stage III-oligometastatic stage IV melanoma, and to find effective biomarkers of efficacy based on tumor paraffin tissue specimens and peripheral blood.

The main questions it aims to answer are:

* The efficacy and safety of the combination treatment regimen;
* Finding suitable biomarkers can refine the patients with effective treatment

After a series of evaluation, if the participants meet the inclusion and exclusion criteria and are evaluated by the investigator, they will formally enter the study observation period and receive the following treatments Endostar: The dose of 210 mg (14 vials) is administered by intravenous pump from Day 1 to Day 3 of each course, every 4 weeks as a cycle, until disease recurrence, metastasis or intolerable toxicity, and up to 6 courses of administration.

Toripalimab: 3 mg/kg by intravenous drip every 2 weeks (Day 1 and Day 15 of each cycle) in a 4-week cycle until disease recurrence, metastasis, or intolerable toxicity for up to 1 year (about 13 cycles).

ELIGIBILITY:
Inclusion Criteria:

1. 18 Age ≤ age ≤75 years old;
2. ECOG performance status: 0 - 1 score;
3. Patients with malignant melanoma confirmed by pathology and/or cytology, except mucosal malignant melanoma and uveal malignant melanoma;
4. Patients who have not received anti-tumor therapy at the initial stage of treatment;
5. Patients with stage III or oligometastasis stage IV malignant melanoma confirmed by histopathology or cytology. Stage III is defined as at least one clinically accessible lymph node metastasis; oligometastasis stage IV is defined as less than 4 metastases and the site of metastasis excludes bone metastases, brain metastases, or other metastases that cannot be completely surgically treated;
6. Complete surgical resection within 13 weeks prior to enrollment;
7. Laboratory tests are required to meet:

   1. Blood routine examination: hemoglobin (Hb) ≥90g/L (no blood transfusion within 14 days); Absolute neutrophil count (NEUT) ≥1.5×109/L; Platelet (PLT) ≥100×109/L;
   2. Biochemical examination: alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5×ULN; Serum total bilirubin (TBIL) ≤1.5×ULN; Serum creatinine (Cr) ≤1.5×ULN and creatinine clearance 50μmol/L;
   3. Coagulation function: activated partial thromboplastin time (APTT), international normalized ratio (INR), prothrombin time (PT) ≤1.5×ULN;
   4. Doppler ultrasound assessment: left ventricular ejection fraction (LVEF)≥50%;
8. Women should agree that they must use contraception (e.g., intrauterine device [IUD], birth control pills, or condoms) during the study and for 6 months after the end of the study; A negative serum or urine pregnancy test within 7 days prior to study enrollment and must be non-lactating; Men should agree to use contraception during the study and for 6 months after the end of the study period;
9. Patients voluntarily joined the study, signed informed consent, and had good compliance and were able to be followed up by the trial staff.

Exclusion Criteria:

1. Patients with a history of allergic reactions to biological products;
2. Patients with previous or concurrent malignancies within 5 years (except for cured basal cell carcinoma of the skin and carcinoma in situ of the cervix);
3. Any active autoimmune disease or history of autoimmune disease (such as, but not limited to, Autoimmune hepatitis, interstitial pneumonia, enteritis, Vasculitis, nephritis; asthma in which the subject needs medical intervention with Bronchiectasis cannot be included); However, the following patients are allowed to be included: Vitiligo, psoriasis, alopecia without systemic treatment, well controlled type I diabetes, hypothyroidism with normal thyroid function after replacement treatment;
4. Patients who need to use immunosuppressants, or systemic or absorbable local hormone therapy to achieve immunosuppression (dose>10mg/day prednisone or other equivalent therapeutic hormone), and continue to use within 2 weeks after the first administration;
5. Patients with any signs or history of bleeding, regardless of severity; Patients with any bleeding or bleeding event ≥CTCAE Grade 3 within 4 weeks prior to the first dose; Or digestive tract diseases such as unhealed wound, fracture, active gastric and duodenal ulcer, ulcerative colitis or active bleeding of unresected tumor, or other conditions that may cause gastrointestinal bleeding and perforation as judged by the investigator;
6. Patients with any severe and/or uncontrolled disease, including:

   1. Patients with poorly controlled blood pressure (systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥90mmHg);
   2. Unstable angina pectoris, myocardial infarction, ≥ Grade 2 congestive heart failure, or arrhythmia requiring treatment (including QTc≥480ms) within 6 months after the first administration;
   3. Active or uncontrolled serious infection (≥CTCAE 2);
   4. Known history of clinically significant liver disease, including viral hepatitis, and known hepatitis B virus (HBV) carriers must exclude active HBV infection, i.e., HBV DNA positive (>1×103 copies/mL or>500 IU/mL); Known hepatitis C virus (HCV) infection and HCV RNA positive (>1×1000 copies/mL or>100 IU/mL), or other decompensated liver disease, chronic hepatitis requiring antiviral therapy;
   5. HIV test positive;
   6. Diabetes mellitus poorly controlled (fasting blood glucose ≥CTCAE 2);
   7. Urine routine examination indicates urine protein ≥++, and 24-hour urine protein quantification is confirmed to be>1.0 g;
7. According to the judgment of the investigator, the patient has other factors that may lead to the forced termination of the study, such as other serious diseases (including mental diseases) requiring concomitant treatment, serious laboratory abnormalities, family or social factors that may affect the safety of the subject, or the collection of data and samples.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
RFS | One year after the first intravenous drip
  recurrence-free survival

SECONDARY OUTCOMES:
DMFS | One year after the first intravenous drip
  Distant metastasis-free survival
OS | One year after the first intravenous drip
  Overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No